CLINICAL TRIAL: NCT01937104
Title: Comparison of Optic Nerve Sheath Diameter According to Position During Laparoscopy
Brief Title: ONSD According to the Position During Laparoscopy
Acronym: ONSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Jung, Assist professor, Chosun University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONSD-P
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Cholecystitis; Ovarian Cyst; Ovarian Cancer; Uterine Myoma; Cervical Cancer
Keywords: Intracranial pressure; Laparoscopy; Optic nerve sheath diameter; Position
MeSH Terms: conditions — Cholecystitis; Ovarian Cysts; Ovarian Neoplasms; Myofibroma; Uterine Cervical Neoplasms | interventions — Desflurane; Remifentanil; Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Drug: Desflurane Anesthesia with desflurane in both Group 1 and Group 2 - adjust minimum alveolar concentration (MAC) to maintain bispectral index (BIS) between 40-60
  Drug: Remifentanil Adjuvant continuous administration
  - adjust effect site concentration to maintain changes of vital sign below 20%
  Device: Ultrasonographic measurement of ONSD
  Procedure/Surgery: Mechanical ventilation Maintain the end-tidal carbon dioxide partial pressure between 35 and 40 mmHg and peak inspiratory pressure below 30 cmH2O.
  Trendelenburg position - 30 degree
  Interventions: Drug: Desflurane; Drug: Remifentanil; Device: Ultrasonographic measurement of ONSD; Procedure: Mechanical ventilation; Procedure: Trendelenburg position - 30 degree
- Group 2 (Experimental): Drug: Desflurane Anesthesia with desflurane in both Group 1 and Group 2 - adjust MAC to maintain BIS between 40-60
  Drug: Remifentanil Adjuvant continuous administration
  - adjust effect site concentration to maintain changes of vital sign below 20%
  Device: Ultrasonographic measurement of ONSD
  Procedure/Surgery: Mechanical ventilation Maintain the end-tidal carbon dioxide partial pressure between 35 and 40 mmHg and peak inspiratory pressure below 30 cmH2O.
  Reverse Trendelenburg position - 30 degree
  Interventions: Drug: Desflurane; Drug: Remifentanil; Device: Ultrasonographic measurement of ONSD; Procedure: Mechanical ventilation; Procedure: Reverse Trendelenburg position - 30 degree

INTERVENTIONS:
Drug: Desflurane — Anesthesia with desflurane in both Group 1 and Group 2
  - adjust MAC to maintain BIS between 40-60
Drug: Remifentanil — Adjuvant continuous administration
  - adjust effect site concentration to maintain changes of vital sign below 20%
  Other Names: Ultiva
Device: Ultrasonographic measurement of ONSD — Patients were placed in the supine position with their eyes closed, and a thick gel layer was applied to the closed upper eyelid. The 7.5-MHz linear probe was placed on the gel without excessive pressure and adjusted to the proper angle for displaying the entry of the optic nerve into the globe. The intensity of the ultrasound was adjusted to display optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band. An ultrasound beam was focused on the retrobulbar area (4 cm deep) using the lowest possible acoustic power that could measure ONSD. The ONSD was measured 3 mm behind the optic disc. Measurements were performed in the transverse and sagittal planes of both eyes, and the final ONSD value was calculated by averaging 4 measured values.
Procedure: Mechanical ventilation — After tracheal intubation, the lungs of the patients were then ventilated with oxygen in air (1:2) using a tidal volume of 8-10 mL/kg and a respiratory rate of 10-12/min, and the ventilation rate was adjusted to maintain the end-tidal carbon dioxide partial pressure between 35 and 40 mmHg and peak inspiratory pressure below 30 cmH2O.
Procedure: Trendelenburg position - 30 degree — Trendelenburg position - 30 degree
  Arms: Group 1
Procedure: Reverse Trendelenburg position - 30 degree — Reverse Trendelenburg position - 30 degree
  Arms: Group 2

SUMMARY:
Increase of intracerebral pressure (ICP) during laparoscopic surgery has known to be associated with positional changes. Optic nerve sheath diameter (ONSD) has correlation with ICP and ultrasonographic measurement of optic nerve sheath diameter (ONSD) is known to be a noninvasive and rapidly applicable technique for evaluating ICP. The aim of this study is to investigate the change of ONSD according to the positional change during laparoscopic surgery.

DETAILED DESCRIPTION:
1. Purpose There can be many physiologic changes during laparoscopic surgery. Increase of intracerebral pressure (ICP) is one of them, which has known to be associated with arterial concentration of carbon dioxide or positional changes. Changes of ICP can be measured directly by invasive method. However, optic nerve sheath diameter (ONSD) has correlation with ICP and ultrasonographic measurement of optic nerve sheath diameter (ONSD) is known to be a noninvasive and rapidly applicable technique for evaluating ICP. The aim of this study is to investigate the change of ONSD according to the positional change during laparoscopic surgery.
2. Hypothesis Changes of ONSD will be shown according to the positional change during laparoscopic surgery, and these can reflect the changes of ICP.
3. Objectives Female patients who are scheduled to undergo laparoscopic surgery, American society of anesthesiologist class (ASA) I-II, aged between 19 to 65 years, are allocated into 2 groups.

   * Group 1: Laparoscopic gynecological surgery, (Trendelenburg position)
   * Group 2: Laparoscopic cholecystectomy, (Reverse trendelenburg position)
4. Methods Patients are premedicated with midazolam 0.5 mg/kg before transported to the operating room. Once in the operating room, patients were monitored with electrocardiography, non invasive blood pressure, pulse oximetry (Datex-Ohmeda S/5, Planar Systems, Inc., Beaverton, OR, USA) and BIS (Aspect 2000, Aspect Medical Systems, Inc., Newton, MA, USA).

   Anesthesia are induced with propofol (2mg/kg) and followed by administering rocuronium 0.6 mg/kg. After tracheal intubation, the lungs of the patients were then ventilated with oxygen in air (1:2) using a tidal volume of 8-10 mL/kg and a respiratory rate of 10-12/min, and the ventilation rate was adjusted to maintain the end-tidal carbon dioxide partial pressure between 35 and 40 mmHg and peak inspiratory pressure below 30 cmH2O. Anesthesia is maintained with desflurane in addition to the continuous infusion of remifentanil. Radial arterial cannulation is done for invasive arterial blood pressure monitoring.

   After induction of anesthesia, when stabilization of cardiovascular status is achieved, optic nerve sheath diameter (ONSD) is measured by ultrasonographic measurement. Patients were placed in the supine position with their eyes closed, and a thick gel layer was applied to the closed upper eyelid. The 7.5-MHz linear probe was placed on the gel without excessive pressure and adjusted to the proper angle for displaying the entry of the optic nerve into the globe. The intensity of the ultrasound was adjusted to display optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band. An ultrasound beam was focused on the retrobulbar area (4 cm deep) using the lowest possible acoustic power that could measure ONSD. The ONSD was measured 3 mm behind the optic disc. Measurements were performed in the transverse and sagittal planes of both eyes, and the final ONSD value was calculated by averaging 4 measured values.

   ONSD was measured at 7 serial time points during surgery:
   1. Preinduction (prior to the induction of anesthesia in the operating room)
   2. 5 minutes after induction of anesthesia
   3. 5 minutes after introducing pneumoperitoneum
   4. 5 minutes after positional change
   5. 15 minutes after positional change
   6. 30 minutes after positional change
   7. 5 minutes after discontinuing pneumoperitoneum Arterial blood gas analysis is performed to evaluate the arterial carbon dioxide concentration (PaCO2) level at each time point.
5. Statistical Analysis All data are expressed as numbers (%) or mean ± standard deviation. Repeated measures ANOVA will be performed to compare the parameters at specific time points during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are scheduled to undergo laparoscopic surgery, American society of anesthesiologist class (ASA) I-II, aged between 19 to 65 years

Exclusion Criteria:

* Aged unger 18 years or over 65 years
* American society of anesthesiologist class (ASA) III-IV
* Patients with increased intracranial pressure (e.g. hydrocephalus, intracranial hemorrhage, etc.)
* Patients with opthalmologic disease

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
ONSD and PaCO2 | 5 minutes after introducing positional change
  ONSD and PaCO2 - 5 minutes after introducing positional change

SECONDARY OUTCOMES:
ONSD and PaCO2 | 5 minutes after introducing pneumoperitoneum
  ONSD and PaCO2 - 5 minutes after introducing pneumoperitoneum

OTHER OUTCOMES:
Preinduction ONSD | prior to the induction of anesthesia, an expected average of 5 minutes
  ONSD - preinduction (prior to the induction of anesthesia in the operating room)
ONSD and PaCO2 | 5 minutes after induction of anesthesia
  ONSD and PaCO2 - 5 minutes after induction of anesthesia
ONSD and PaCO2 | 15 minutes after positional change
  ONSD and PaCO2 - 15 min after positional change
ONSD and PaCO2 | 30 minutes after positional change
  ONSD and PaCO2 - 30 minutes after positional change
ONSD and PaCO2 | 5 minutes after discontinuing pneumoperitoneum
  ONSD and PaCO2 - 5 minutes after discontinuing pneumoperitoneum

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Jung, M.D., Study Chair — Department of Anesthesiology and Pain medicine School of Medicine, Chosun University
Locations (1):
- Chosun University Hospital, Gwangju, Donggu, South Korea

REFERENCES:
- [Result] Gerges FJ, Kanazi GE, Jabbour-Khoury SI. Anesthesia for laparoscopy: a review. J Clin Anesth. 2006 Feb;18(1):67-78. doi: 10.1016/j.jclinane.2005.01.013. PMID 16517337
- [Result] Moretti R, Pizzi B. Ultrasonography of the optic nerve in neurocritically ill patients. Acta Anaesthesiol Scand. 2011 Jul;55(6):644-52. doi: 10.1111/j.1399-6576.2011.02432.x. Epub 2011 Apr 4. PMID 21463263
- [Result] Geeraerts T, Newcombe VF, Coles JP, Abate MG, Perkes IE, Hutchinson PJ, Outtrim JG, Chatfield DA, Menon DK. Use of T2-weighted magnetic resonance imaging of the optic nerve sheath to detect raised intracranial pressure. Crit Care. 2008;12(5):R114. doi: 10.1186/cc7006. Epub 2008 Sep 11. PMID 18786243
- [Result] Moretti R, Pizzi B, Cassini F, Vivaldi N. Reliability of optic nerve ultrasound for the evaluation of patients with spontaneous intracranial hemorrhage. Neurocrit Care. 2009 Dec;11(3):406-10. doi: 10.1007/s12028-009-9250-8. PMID 19636971
- [Result] Geeraerts T, Launey Y, Martin L, Pottecher J, Vigue B, Duranteau J, Benhamou D. Ultrasonography of the optic nerve sheath may be useful for detecting raised intracranial pressure after severe brain injury. Intensive Care Med. 2007 Oct;33(10):1704-11. doi: 10.1007/s00134-007-0797-6. Epub 2007 Aug 1. PMID 17668184